CLINICAL TRIAL: NCT06137820
Title: Randomized Placebo-controlled Multi-center Study of Efficacy and Safety of a CFA-based Topical Cream Cetilar®️ in Patients With Ankle Injury or Chronic Trauma to the Ankle
Brief Title: CETI-ANKLE: Cetilar®️ in Patients With Ankle Injury or Chronic Trauma to the Ankle
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Pharmanutra S.p.a. (Industry)
Collaborators: NEA Clinical S.r.l. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CET 01/22
Record Dates: First submitted 2023-10-18; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Ankle Injury or Chronic Trauma to the Ankle
Keywords: Ankle injury; Chronic trauma; Ankle trauma; Cetilar
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Cetilar®) (Experimental): Participants received Cetilar® topical cream twice daily for 30 days. An average amount of 5 g per day
  Interventions: Device: Cetilar® (topical cream)
- Control group (Placebo) (Placebo Comparator): Participants received Cetilar Placebo topical cream twice daily for 30 days. An average amount of 5 g per day
  Interventions: Device: Cetilar Placebo

INTERVENTIONS:
Device: Cetilar® (topical cream) — Topical cream twice daily for 30 days. An average amount of 5 g per day.
  Arms: Treatment group (Cetilar®)
Device: Cetilar Placebo — Cetilar placebo cream matching to Cetilar®. Topical cream twice daily for 30 days. An average amount of 5 g per day
  Arms: Control group (Placebo)

SUMMARY:
The purpose of this study is to assess the safety, tolerability and efficacy of Cetilar®

DETAILED DESCRIPTION:
After being informed about the study, all patients giving written informed consent will undergo no more than a 1-week screening period to determine eligibility for study entry. Patients that meet inclusion criteria and do not have exclusion criteria will be randomized in a double-blind manner (participant and investigator) in a 1:1 ratio to Cetilar® cream (about 5 g, twice per day) or placebo cream (about 5 g, twice per day).

ELIGIBILITY:
Inclusion Criteria:

1. Signing the Patient Information Sheet and Informed Consent Form
2. Patients with reduced ankle mobility caused by injury or chronic trauma to the ankle
3. Men or women aged ≥20 and ≤80 years
4. Patients who mark the pain 4 cm on a VAS
5. Patients who are willing or able to follow doctor's instructions
6. Patients not participating in other clinical trials within 30 days before the screening
7. Patients who have received sufficient explanation for this clinical trial and agreed to participate

Exclusion Criteria:

1. Patients who received intraarticular injection treatment into the painful area within 3 months prior to the first visit
2. Ankle surgery in the previous six months
3. Topical NSAIDs application during the treatment period
4. BMI > 32
5. Systemic inflammatory diseases (e.g. fibromyalgia, etc.)
6. Progressive serious medical conditions (such as cancer, AIDS or end-stage renal disease)
7. Patients with major infections in the observation period
8. Renal diseases (serum creatinine concentration more than 1.2 times the upper limit of the normal range according to the central laboratory definition reference values)
9. Liver dysfunction (serum alanine or aspartate transaminase concentrations more than 1.5 times the upper limit of normal range)
10. Patients with serious heart-related diseases such as cardiac arrest, a history of cerebral infarction, or ischemic heart disease
11. Patients who received systemic steroid treatment within 1 month prior to their first visit
12. Diabetic foot
13. Pregnant or lactating women

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-11-18 (Actual); Primary Completion 2023-08-19 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in FAAM (Foot and Ankle Ability and Measure) total score questionnaire on day 30 | From Baseline to Day 30
  FAAM is a validated questionnaire assessing mobility and functionality on Day 30. Change = (Day 30 - Baseline Score).
  This instrument includes 2 subscales:
  1. Activities of Daily Living (ADLs) subscale of 21 items
  2. Sports subscale of 7 items. For each subscale patients were asked to answer each question with a single response that most clearly described their condition within the past week.
  Answers for both scales are based on a Likert scale (4-0) of:
  4) "no difficulty" 3) "slight difficulty" 2) "moderate difficulty"
  1) "extreme difficulty" 0) "unable to do" If an activity in question was limited by something other than their ankle, the patient was asked to record N/A To calculate the score for either subscale, the total number of points are added, divided by the total number of possible and then multiplied by 100.
  Therefore, a higher score reflects a higher level of physical function.
Change From Baseline in Pain on the Visual Analogue Scale (VAS scale) on day 30 | From Baseline to Day 30
  Visual analogue scale (VAS) is a validated questionnaire assessing pain intensity on Day 30. Possible scores range from 0 cm (no pain) to 10 cm (Pain as bad as it could be). Change = (Day 30 - Baseline Score).
Change From Baseline in QoL (Quality of Life) total score questionnaire on day 30 | From Baseline to Day 30
  QoL is a validated questionnaire assessing taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, general mental health, social functioning, energy/fatigue, and general health perceptions on Day 30. Change = (Day 30 - Baseline Score). Scale scores represent the average for all items in the scale that the patients answered.

SECONDARY OUTCOMES:
The number and % of patients with treatment-emergent adverse events | From Baseline to Day 30
  Incidence and severity of adverse events (AEs) that occurred during the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Sole Rossato, Study Director — Pharmanutra S.p.a.
Locations (3):
- Georgia (2):
  - LLC "Altra Vita", Tbilisi
  - JSC "Evex Hospitals" (Caraps Medline), Tbilisi
- Azienda Sanitaria Locale Viterbo | ASL Viterbo, Dipartimento di Ortopedia (Centro Coordinatore), Viterbo, Italy

IPD SHARING:
Plan to Share IPD: No